CLINICAL TRIAL: NCT06524804
Title: A Phase Ib/II Clinical Study Evaluating the Safety, Tolerability, Efficacy, and Pharmacokinetic Characteristics of BY101298 Combined with Radiotherapy in Patients with Malignant Solid Tumors
Brief Title: A Phase Ib/II Study of BY101298 , an Oral DNA-PK Inhibitor, Combined with Radiotherapy in Patients with Malignant Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The sponsor adjusts the clinical development strategy.
Sponsor: Chengdu Baiyu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BY1298-I-02
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-05

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BY101298 in combination with palliative radiotherapy (Experimental): Patients in Phase I undergo palliative radiotherapy for 5 fractions per week and receive BY101298 PO QD concomitant with radiation therapy.
  Interventions: Drug: BY101298 Capsules; Radiation: palliative radiotherapy
- BY101298 in combination with curative radiotherapy (Experimental): Patients in Phase I undergo curative radiotherapy for 5 fractions per week and receive BY101298 PO QD concomitant with radiation therapy.
  Interventions: Drug: BY101298 Capsules; Radiation: curative radiotherapy

INTERVENTIONS:
Drug: BY101298 Capsules — An oral DNA-PK Inhibitor
  Arms: BY101298 in combination with palliative radiotherapy
Radiation: palliative radiotherapy — Undergo palliative radiotherapy
  Arms: BY101298 in combination with palliative radiotherapy
Drug: BY101298 Capsules — An oral DNA-PK Inhibitor
  Arms: BY101298 in combination with curative radiotherapy
Radiation: curative radiotherapy — Undergo curative radiotherapy
  Arms: BY101298 in combination with curative radiotherapy

SUMMARY:
BY101298 is an innovative DNA-dependent protein kinases (DNA-PK) highly selective small molecule inhibitor. DNA-dependent protein kinases (DNA-PK plays a key role in the NHEJ repair pathway to repair DNA double-strand breaks (DSBs). By inhibiting DNA-PK activity to inhibit DSBs repair, BY101298 may synergistically improve the killing effect on tumor cells, reduce the risk of local recurrence and metastasis, and improve the clinical benefit of cancer patients when combing with radiotherapy.

Primary objective is to assess the safety and tolerability; RP2D. The secondary Objectives are to characterize the pharmacokinetic (PK) profile of BY101298 and to assess the preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, ≥ 18 and ≤ 75 years of age (inclusive at the time of informed consent).
2. histologically or cytologically diagnosed solid tumors with indications for radiotherapy after evaluation by investigator (Radiotherapy sites are excluded for patients with primary brain tumors and/or brain metastases). Radiotherapy techniques could be IMRT, IGRT, VMAT or TOMO, except SBRT and SRS.
3. Cohort 1: Patients with locally advanced/advanced malignant solid tumors who will receive radiotherapy for non-radical purposes, such as radiotherapy for non-oligometastatic tumors.
4. Cohort 2: Radiotherapy for radical purposes [including, but not limited to, radiotherapy for residual or oligofocal lesions with stable disease or partial response (SD, PR) after systemic treatment, sequential chemoradiotherapy, or not suitable for chemotherapy] with at least one measurable lesion present in the radiation field according to RECIST 1.1 criteria, and radiotherapy dose following each solid tumor radiotherapy guideline. The segmentation method is conventional segmentation.
5. After obtaining RP2D doses in Phase Ib, extended studies were conducted in specific indications in cohort 1 and Cohort 2, respectively.
6. Life expectancy ≥ 3 months (cohort 1), and ≥ 6 months (cohort 2).
7. The lesions outside the radiation field are tended to be stabilized evaluated by the investigator.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 1. (If the symptoms are caused by tumor lesions in the radiotherapy field, ECOG score 0-2 points).
9. Adequate organ and bone marrow function. Laboratory tests that meet the following criteria within 7 days prior to the first dose of study treatment (without blood transfusion, erythropoietin, recombinant human thrombopoietin or colony stimulating factor therapy, renal replacement therapy, etc., within 14 days prior to the screening examination).
10. Understand and be willing to sign written informed consent and be able to follow the study protocol for treatment, visits, and other study procedures.

Exclusion Criteria:

1. Treated with DNA-PK inhibitors.
2. Potential risks of perforation, bleeding, or other unacceptable risks after treatment evaluated by the investigator.
3. Radiotherapy sites are primary brain tumors and/or brain metastases.
4. Previous treatment with any of the following:

   1. Patients who have received systemic chemotherapy, traditional Chinese medicine for anti-tumor indications or other anti-tumor drugs (including endocrine therapy, molecular targeted therapy, immunotherapy, biological therapy, etc.) within 4 weeks or 5 half-lives (whichever is longer) prior to the first dose of the study drug, or those who need to continue receiving these drugs during the study.
   2. Received radiation therapy in the planned radiotherapy field (re-course and multi-course same-site radiotherapy should be excluded in principle).
   3. The patient has previously received radiotherapy at another site, unless there is no potential risk based on OAR exposure evaluated by the investigator.
   4. Received chinese troditional medicine (Chinese patent medicine) with antitumor indications within 2 weeks prior to initial administration of the investigational drug.
5. Major surgery (craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to the first dose of the study drug and surgery is scheduled during the study period.
6. Brain metastasis (except asymptomatic, stable for more than 4 weeks prior to the first dose and not requiring steroid therapy for at least 4 weeks prior to the first dose, no imaging findings of marked edema around the tumor lesion), presence of meningeal metastasis or brainstem metastasis, or presence of spinal cord compression.
7. Concomitant with other malignancies that may affect the patient's expected life expectancy.
8. Have undergone bone marrow transplants and/or organ transplants, including allogeneic stem cell transplants.
9. Toxicities from prior antitumor therapy that have not recovered to CTCAE version 5.0 Grade 1 or less, except CTCAE (V5.0) Grade 2 peripheral neurotoxicity and alopecia of any grade, and other toxicity that has no safety risk evaluated by the investigator.
10. Patients with third lacunar effusion (such as large pleural effusion, ascites, or pericardial effusion) which is difficult to control and requires repeated drainage.
11. Serious or uncontrolled diseases as assessed by the investigator, including but not limited to:

    1. Severe or uncontrolled diabetes (fasting blood glucose ≥ 10 mmol/L), poorly controlled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg under standardized antihypertensive regimens), epilepsy, chronic obstructive pulmonary disease, interstitial pneumonia, pulmonary interstitial fibrosis, Parkinson 's disease, active bleeding, uncontrolled infection.
    2. Cognitive dysfunction, history of psychiatric disorders, other uncontrolled concomitant diseases, alcohol dependence, hormone dependence, or drug abuse.
    3. History of immunodeficiency, including HIV antibody positive, other acquired or congenital immunodeficiency disease, or history of organ transplantation.
    4. HBsAg or HBcAb positive, and peripheral blood HBV DNA titer test ≥ 200 IU/mL or ≥ 1000 copies/mL or above the upper limit of normal value at the study site; HCV antibody test positive, and HCV RNA test above the upper limit of normal value at the study site; treponema pallidum-specific antibody positive.
    5. Clinically serious gastrointestinal dysfunction that may compromise drug intake, transport, or absorption. For example, inability to take oral medication, uncontrollable nausea or vomiting, history of massive gastrointestinal resection, history of gastrointestinal ulcer and gastrointestinal bleeding within 6 months prior to the first dose, untreated recurrent diarrhea, untreated stomach disease requiring long-term use of PPI acid suppressants, Crohn 's disease, ulcerative colitis, etc.
    6. Prior thyroid dysfunction or inability to maintain thyroid function within normal limits even with medical therapy.
12. Cardiac dysfunction, including any of the following:

    1. Myocardial infarction in past 6 months, heart failure classified as Class II/III/IV according to the New York Heart Association (NYHA) Functional Classification, unstable angina pectoris, and unstable arrhythmia.
    2. Left ventricular ejection fraction LVEF < 50% shown by echocardiography.
    3. QT interval corrected using Fridericia 's formula: QTcF > 470 msec (females), QTcF > 450 msec (males).
13. Pregnant (positive pregnancy test prior to dosing) or lactating.
14. History of serious hypersensitivity (e.g., anaphylactic shock) or hypersensitivity to excipients or other ingredients associated with the study drug.
15. Received live attenuated vaccine within 28 days prior to the first dose.
16. Other factors considered unsuitable for study enrollment by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of BY101298 combined with radiotherapy in patients with advanced malignant solid tumors. | through study completion (an average of 1.5 years)
  Grade and frequency of adverse events and serious adverse events
To assess the maximum tolerated dose (MTD) | through study completion (an average of 1.5 years)
  Incidence of Dose limiting Toxicities (DLTs)
To determine the recommended phase II dose of BY101298 combined with radiotherapy in patients with advanced malignant solid tumors. | through study completion (an average of 1.5 years)
  the recommended phase II dose（RP2D）

SECONDARY OUTCOMES:
To evaluate the pharmacokinetic (PK) characteristics of BY101298 combined with radiotherapy in patients with advanced malignant solid tumors. | through study completion (an average of 1.5 years)
  AUC
To evaluate the pharmacokinetic (PK) characteristics of BY101298 combined with radiotherapy in patients with advanced malignant solid tumors. | through study completion (an average of 1.5 years)
  Cmax
To evaluate the pharmacokinetic (PK) characteristics of BY101298 combined with radiotherapy in patients with advanced malignant solid tumors. | through study completion (an average of 1.5 years)
  Cmax,ss
To evaluate the pharmacokinetic (PK) characteristics of BY101298 combined with radiotherapy in patients with advanced malignant solid tumors. | through study completion (an average of 1.5 years)
  Cmin,ss
To evaluate the preliminary efficacy of BY101298 combined with radiotherapy in patients advanced malignant solid tumors. | through study completion (an average of 1.5 years)
  ORR
To evaluate the preliminary efficacy of BY101298 combined with radiotherapy in patients advanced malignant solid tumors. | through study completion (an average of 1.5 years)
  DCR
To evaluate the preliminary efficacy of BY101298 combined with radiotherapy in patients advanced malignant solid tumors. | through study completion (an average of 1.5 years)
  DOR
To evaluate the preliminary efficacy of BY101298 combined with radiotherapy in patients advanced malignant solid tumors. | through study completion (an average of 1.5 years)
  PFS
To evaluate the preliminary efficacy of BY101298 combined with radiotherapy in patients advanced malignant solid tumors. | through study completion (an average of 1.5 years)
  OS

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Affiliated to Shandong First Medical University / Shandong Cancer Research Institute / Shandong Cancer Hospital, Jinan, Shandong, China